CLINICAL TRIAL: NCT06909383
Title: Nanocrystalline Megestrol Acetate for the Treatment of Anorexia-Cachexia Syndrome in Extensive-Stage Small Cell Lung Cancer: A Prospective, Open-Label, Single-Arm Phase II Clinical Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Zhou Chengzhi, Vice President of the First Affiliated Hospital of Guangzhou Medical University, Guangzhou Institute of Respiratory Disease
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CROC-25-01
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Extensive-stage Small Cell Lung Cancer (ES-SCLC); Cancer - Associated Anorexia - Cachexia Syndrome
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Nanocrystalline megestrol acetate+immunochemotherapy (Experimental)
  Interventions: Drug: Nanocrystalline megestrol acetate

INTERVENTIONS:
Drug: Nanocrystalline megestrol acetate — Nanocrystalline megestrol acetate

SUMMARY:
Patients with extensive-stage small cell lung cancer are a high-risk group for cancer cachexia and anorexia. Meanwhile, the adverse reactions of chemotherapy and immunotherapy potentially exacerbate the occurrence and development of cancer cachexia and anorexia. Cancer cachexia and anorexia also severely affect the quality of life of patients with extensive-stage small cell lung cancer, significantly shortening their overall survival (OS) and progression-free survival (PFS), thus forming a vicious cycle.

Numerous previous studies have shown that for patients with advanced tumors, the combination of supportive treatments such as megestrol acetate during chemotherapy or concurrent chemoradiotherapy is a treatment mode with clinical significance and practical feasibility in clinical practice. However, the efficacy and the optimal treatment timing of its combination with the current first-line immunochemotherapy regimen remain unclear. Although mechanistic studies have shown that anti-cachexia treatment may synergistically enhance the efficacy of immunotherapy, there is a lack of relevant clinical research evidence.

ELIGIBILITY:
Inclusion Criteria:

Patients who have been confirmed by histological or cytological examination to have small cell lung cancer (SCLC), and who have been identified as having extensive-stage small cell lung cancer based on the 8th edition of the AJCC staging system or the Veterans Administration Lung Group (VALG) criteria (excluding patients with combined small cell lung cancer).

The subjects have not received systemic chemotherapy for metastatic diseases in the past. For subjects who have previously received adjuvant/neoadjuvant chemotherapy aimed at cure for non-metastatic diseases, or radical concurrent or sequential chemoradiotherapy, if the disease progression occurs more than 6 months after the end of the last treatment, they are eligible to participate in this study.

According to RECIST v1.1, there is at least one measurable tumor lesion. Meet the diagnostic criteria for the pre-cachexia or cachexia stage. -

Exclusion Criteria:

1. Cancer-specific exclusion criteria:

   1. Active or untreated CNS metastases (e.g., brain or leptomeningeal metastases) determined by CT or magnetic resonance imaging (MRI) evaluation during screening and previous imaging evaluations. Patients who have previously received treatment for brain or leptomeningeal metastases, have been stable for ≥ 2 months, and have discontinued systemic hormonal therapy (> 10 mg/day of prednisone or equivalent) for > 4 weeks before randomization may participate in the study.
   2. Uncontrolled tumor-related pain;
   3. Thromboembolic disease, ascites, or lower extremity edema within the past 6 months;
   4. A history of malignant tumors other than lung cancer within 5 years before random assignment, except for malignant tumors with a negligible risk of metastasis or death [e.g., with an expected 5-year overall survival rate > 90%] and those expected to be cured after treatment, such as appropriately treated cervical carcinoma in situ, basal or squamous cell skin cancer, localized prostate cancer treated with radical surgery, and ductal carcinoma in situ treated with radical surgery;
   5. Persistent toxicity from previous anti-tumor treatment that has not been resolved. "Not resolved" is defined as not having recovered to grade 0 or 1 according to NCI CTCAE version 5.0 (excluding alopecia) or not having recovered to the level specified in the inclusion/exclusion criteria.
2. General medical exclusion criteria:

   1. Women who are pregnant, lactating, or planning to become pregnant during the study period;
   2. Patients with hepatitis B (known to be positive for HBV surface antigen HBsAg and with HBV DNA detected at each study center ≥ 1000 cps/ml or 200 IU/ml or ≥ the upper limit of the normal value) or hepatitis C:

      * For patients with a previous history of hepatitis B virus (HBV) infection, HBV deoxyribonucleic acid (DNA) testing must be performed on this group of patients. Only those with a negative HBV DNA result (HBV DNA < 1000 cps/ml or 200 IU/ml or below the upper limit of the normal value) are eligible to participate in this study;
      * Among patients with a positive hepatitis C virus (HCV) antibody, only those with a negative polymerase chain reaction (PCR) HCV ribonucleic acid (RNA) result can participate in this study.
   3. Patients with a positive test result for human immunodeficiency virus (HIV);
   4. Those who have undergone major surgery (excluding diagnostic surgery) within 28 days before random assignment, or are expected to undergo major surgery during the study period;
   5. Significant cardiovascular diseases, such as heart diseases defined by the New York Heart Association (Class II or higher), myocardial infarction occurred within 3 months before random assignment, unstable arrhythmia, unstable angina pectoris, cerebrovascular accident or transient ischemic attack; Patients known to have coronary artery disease, congestive heart failure that does not meet the above criteria, or with a left ventricular ejection fraction < 50% must receive the optimal stable treatment regimen considered by the attending physician, and consultation with a cardiologist is advisable if necessary;
   6. Severe infections occurred within 4 weeks before the first administration, including but not limited to those with comorbidities requiring hospitalization, sepsis, or severe pneumonia; Active infections (excluding antiviral treatment for hepatitis B or hepatitis C) for which systemic anti-infective treatment was received within 2 weeks before the first administration.
3. Exclusion criteria related to drug use:

   1. Any condition that affects gastrointestinal absorption, such as dysphagia, malabsorption, uncontrollable vomiting, etc.; Patients with difficulty in food intake or those who require enteral or parenteral nutritional support; Patients with anorexia nervosa, anorexia caused by mental illness, or difficulty in eating due to pain.
   2. Currently taking or planning to take other drugs that increase appetite or body weight, such as adrenal corticosteroids (except for short-term use of dexamethasone during chemotherapy), androgens, progestins, thalidomide, olanzapine, anamorelin, or other appetite stimulants.
   3. Patients with Cushing's syndrome, adrenal or pituitary insufficiency; Patients with poorly controlled diabetes; Patients with current hypertension whose systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg after treatment with oral antihypertensive drugs.
   4. A history of esophageal-gastric varices, severe ulcers, gastrointestinal perforation and/or fistula, a history of gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), intra-abdominal abscess, or acute gastrointestinal bleeding within 6 months before the first administration.
   5. Known allergy to any component of the study drug.
   6. Other situations that the investigator deems unsuitable.

      -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with a body weight increase of more than 5% relative to the baseline | at the 12th week

IPD SHARING:
Plan to Share IPD: Undecided